CLINICAL TRIAL: NCT00752440
Title: Inspiratory Muscle Training in Patients With Autonomic Neuropathic: a Randomized Trial
Brief Title: Inspiratory Muscle Training in Patients With Autonomic Neuropathic
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Organization: Intituto de Cardiologia do Rio Grande do Sul/ Fundação Universitária de Cardiologia, Beatriz Schann
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 3865/06
Record Dates: First submitted 2008-09-12; First posted 2008-09-15 (Estimated); Last update posted 2008-09-16 (Estimated); Status verified 2008-09

CONDITIONS: Diabetes Mellitus; Diabetic Autonomic Neuropathy
Keywords: Diabetes Mellitus; Autonomic Neuropathy; Inspiratory Muscle training
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Neuropathies | interventions — Vital Capacity; Forced Expiratory Volume

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Inspiratory muscle training (IMT) — IMT (30 min 7 times per week, for 8 weeks)
  Other Names: Diabetic autonomic neuropathy;; Inspiratory muscle function testing;; forced vital capacity and forced expiratory volume;; Maximal functional capacity with incremental exercise test;; variability of the heart frequency.

SUMMARY:
This study describes a controlled randomized clinical trial to evaluate the effect of inspiratory muscle training in patients with diabetic autonomic neuropathy.

DETAILED DESCRIPTION:
The diabetic autonomic neuropathy (NAD) is a common complication of diabetes mellitus (DM), both of the type 1 diabetes mellitus (DM1) as of the type 2 diabetes mellitus (DM2). The results of this study, would help to reveal the degree of commitment generated by NAD in respiratory muscle strength, can also enable the development of a new therapeutic approach, such non-pharmacological (respiratory muscle training), with a view to improve the respiratory muscle strength and alleviate the autonomic dysfunction in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic autonomic neuropathy
* Age between 36 and
* 70 years old and signed in informed consent form

Exclusion Criteria:

* Presence of congestive heart failure
* Chronic obstructive pulmonary disease (FEV1 < 70% and/or FEV1%< 80
* Class II or III obesity (body mass index > 35)

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2006-08; Primary Completion 2008-11 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Inspiratory muscle strength | eight

SECONDARY OUTCOMES:
Variability of heart rate | eight

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz D Schann, MD, ScD, Principal Investigator — Institudo de cardiologia de Porto Alegre
Locations (1):
- Institudo de Cardiologia do Rio Grande do Sul, Porto Alegre, RGS, Brazil